CLINICAL TRIAL: NCT00979667
Title: Multicentre, Randomized, Controlled Clinical Trial Comparing Oseltamivir With Placebo And Zanamivir With Control As The First Line Treatment For Human Swine Influenza (H1N1) Infection In Designated Flu Clinics During The Pandemic Influenza in Hong Kong
Brief Title: A Clinical Trial Comparing Oseltamivir With Placebo And Zanamivir With Control As First Line Treatment For Human Swine Influenza Infection
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Decreased Influenza activity; thus decrease/no eligible patient to recruit
Sponsor: Chinese University of Hong Kong (Other)
Collaborators: Food and Health Bureau, Hong Kong (Other Government); Hospital Authority (Ambiguous)
Responsible Party: Prof. Benny Chung Ying ZEE and Dr. Augustine Tsan LAM, The Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CCT2009-CS-6
Record Dates: First submitted 2009-09-17; First posted 2009-09-18 (Estimated); Last update posted 2011-04-11 (Estimated); Status verified 2010-05

CONDITIONS: Upper Respiratory Tract Infection; Influenza
Keywords: Upper respiratory tract infection; Influenza A; Human Swine Influenza
MeSH Terms: conditions — Respiratory Tract Infections; Influenza, Human | interventions — Oseltamivir; Zanamivir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Oseltamivir (Experimental)
  Interventions: Drug: Oseltamivir
- Zanamivir (Experimental)
  Interventions: Drug: Zanamivir
- Placebo of Oseltamivir (Placebo Comparator)
  Interventions: Drug: Placebo of Oseltamivir

INTERVENTIONS:
Drug: Oseltamivir — 75 mg twice daily for 5 days
  Other Names: Tamiflu
  Arms: Oseltamivir
Drug: Zanamivir — 10 mg twice daily for 5 days
  Other Names: Relenza
  Arms: Zanamivir
Drug: Placebo of Oseltamivir — twice daily for 5 days
  Other Names: Tamiflu Placebo
  Arms: Placebo of Oseltamivir

SUMMARY:
To evaluate the efficacy of oseltamivir ,as compared with the placebo arm and zanamivir with its control arm with respect to symptoms duration among patients infected with influenza A (H1N1) virus.

DETAILED DESCRIPTION:
The outbreak of respiratory illnesses in Mexico that began in March 2009 was caused by a swine origin influenza A (H1N1) virus (S-OIV) that had not been recognized previously in pigs or humans. As of 17 May 2009, 39 countries have officially reported 8480 cases of influenza A (H1N1) infection.

The H1N1 influenza A virus appears sensitive to oseltamivir and zanamivir in vitro, but resistant to amantadine and rimantadine. This study is to test the oseltamivir, zanamivir and placebo arms as the first line treatment for human swine influenza infection. Through the study, the investigators may have better understanding about the clinical and, biochemical, virological profiles of oseltamivir/zanamivir on the H1N1 virus, and optimizing the treatment strategy among the Chinese population.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients 18 years or older with body weight >40kg
* Written informed consent
* Presented within 48 hours of onset of influenza-like illness
* Presumptive diagnosis of H1N1 satisfying the following clinical and laboratory criteria:

  * Clinical criteria

    * Fever >38 oC (Infrared Forehead Thermometer will be used to measure the Temporal Artery Temperature under the skin) AND
    * At least one upper respiratory tract infection (cough, running nose, sore throat)
  * Laboratory criteria Positive rapid test result for influenza A (by Influenza Rapid Diagnostic test) within 48 hours of onset of flu-like symptoms

Exclusion Criteria:

* Age below 18 years
* Persons who lack the ability to care for themselves
* Patient with critical condition or already developed severe respiratory distress with hypoxaemia on presentation
* Pregnancy or lactation
* Coexisting liver disease
* Coexisting cardiovascular disease except stable hypertension without complication
* Coexisting chronic pulmonary disease
* Coexisting immuno-compromised medical conditions or on concurrent immunosuppressive therapies
* Renal failure
* Terminal malignancies or terminal end-organ failure with an estimated life-expectancy of less than 3 months
* Known intolerance to oseltamivir or zanamivir
* Known history of significant neurological disorders that can compromise respiratory function or the handling of respiratory secretions or that can increase the risk for aspiration or those
* Subjects who have received oseltamivir as prophylaxis for H1N1 infection
* Subjects who have received any investigational drug within 1 month prior to study entry
* Subjects with a mental condition rendering the subject unable to understand the nature, scope, and possible consequences of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2009-10; Primary Completion 2010-08 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Time to symptoms resolution as reported by the patient | one week

SECONDARY OUTCOMES:
Treatment failure including hospitalization due to disease worsening. | one week
Viral load | one week
Severity of disease as measured by the patient diary and quality of life using SF12v2. | one week

CONTACTS AND LOCATIONS:
Overall Officials: Augustine T. LAM, MBBS, Principal Investigator — Prince of Wales Hospital, Shatin, Hong Kong
Locations (3):
- Shau Kei Wan Jockey Club Clinic, Hong Kong, Hong Kong, China
- Hong Kong (2):
  - Fanling Family Medicine Centre, Hong Kong
  - Sai Ying Pun Jockey Club General Outpatient Clinic, Hong Kong